CLINICAL TRIAL: NCT04676165
Title: Evaluation of a Mobile Application to Enhance Medication Management Following Hospital Discharge
Brief Title: Mobile Application to Enhance Medication Management
Acronym: SAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Robyn Tamblyn, Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-53
Record Dates: First submitted 2020-12-09; First posted 2020-12-19 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-11

CONDITIONS: Medication Adherence; Mobile Application
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, study participants are not blinded to treatment arm allocation, but data analysts are.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAM Group (Experimental): At discharge from hospital, patients (and/or caregivers) will receive access to Smart About Meds (SAM), a medication management mobile application that has been developed by the McGill Clinical and Health Informatics (MCHI) Research Group.
  Interventions: Device: Smart About Meds (SAM)
- Usual Care Group (No Intervention): At discharge from hospital, patients will be provided with a written discharge prescription to be filled at their community pharmacy, and may or may not receive written or verbal instructions about changes made to therapy.

INTERVENTIONS:
Device: Smart About Meds (SAM) — SAM generates a patient-friendly list of prescribed and dispensed medications and offers several features:
  * Drug information: Patient-friendly monographs that describe treatment indications and the harms/benefits of medications.
  * Adherence alerts: Alerts users to non-adherence, such as when they fill prescriptions that were stopped at hospital discharge, don't fill prescribed medications, or buy medications at the incorrect dose.
  * Side-effect checker: Provides a list of side effects associated with individual medications and the patient's overall drug profile.
  * Rate my med: Allows patients to rate medications and describe experiences with a medication. Patients can view ratings given by users.
  * Caregiver connect: Provides patients' caregivers with access to the app.
  * Pharmacy connect: Allows patients to connect with their hospital pharmacist to ask questions regarding their medications and adherence alerts.
  * Other: pill images, daily pill reminders, weekly dosing schedule
  Arms: SAM Group

SUMMARY:
Adverse drug events (ADEs) are a leading cause of death in North America, with over 2 million ADEs causing 100,000 deaths every year and millions in economic costs. The majority of ADEs that occur within 30 days of discharge from hospital are related to prescription medications and of these, more than 50% are preventable. Among the causes of ADEs are incomplete and unclear medication lists, and a lack of patient understanding and adherence. Patients are usually discharged from hospital on substantially difference medication regiments than those prior to admission. In the absence of supportive mechanisms that ensure patients' understanding of their medication list, adherence to prescribed medication changes is likely to be reduced and the subsequent risk of ADEs increased. Secondary analyses from a recently conducted randomized controlled trial (RCT) by our team suggest that more than 50% of study patient were non-adherent to at least one in-hospital medication change, and that this non-adherence significantly increased the risk of hospital re-admission and emergency department visits in the 30 days post-discharge. Furthermore, analyses of interview data suggest that non-adherence may be driven by unclear communication with patients about medication changes and the reasons for these changes, as well as difficulties in managing complex dosing schedules and drug regimen information. There is therefore a clear need to implement and evaluate patient support mechanisms that reduce non-adherence to essential changes in therapy following hospitalization.

The objective of this project is to conduct a pilot RCT that will evaluate the usability of a medication management mobile application and its efficacy in reducing non-adherence to in-hospital medication changes following discharge. We will randomize 100 patients from the internal medicine unit of the McGill University Health Centre (MUHC) Glen site to either the intervention or control arm. Patients in the control arm will receive usual care (i.e. no medication management support), whereas those in the intervention arm will receive a tablet with the installed mobile application. The application will integrate prescription claims data from the Régie de l'assurance maladie du Québec (RAMQ) for the 3-month period prior to hospital admission with the patient's discharge prescription to generate a patient-friendly medication list, along with details of in-hospital medication changes. The app will also offer a number of features designed to maximize patient understanding and adherence, including pill images, patient-friendly drug monographs, weekly dosing schedules, drug alerts, home refill services, and features that connect with the patient's caregiver and hospital pharmacist.

At 1 week post-discharge, study coordinators will conduct a usability assessment to obtain patient feedback on the app (via a technology acceptance questionnaire) and to document usability using the "think aloud" protocol, which is based on observing and recording patients as they use the application and verbalize any thoughts that might occur to them. Qualitative analysis of recorded and transcribed sessions will then be used to assess the technology's ease of use, user-friendliness, efficiency, and any features that may cause confusion, frustration, or user errors.

Non-adherence to in-hospital treatment changes will be assessed by comparing patients' discharge prescriptions with medications dispensed in the 30 days following hospital discharge (obtained from RAMQ pharmacy claims). We will compare, between intervention and control groups, the average number of in-hospital medication changes not adhered to in the 30-day follow-up period.

This project will assess a technological intervention that has the potential to improve patient adherence to in-hospital medication changes and may subsequently reduce the occurrence of ADEs. Given the high costs associated with ADEs, this small investment has the potential to incur significant cost savings for the Quebec healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Discharged home from internal medicine units of the McGill University Health Center
* Have a mobile or tablet device with internet connection
* Have prescription drug insurance from the provincial health insurer
* Prescribed at least one medication at discharge from hospital

Exclusion Criteria:

* Discharged to a rehabilitation center
* Transferred to a non-study unit'
* Prognosis of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Tamblyn, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University Health Centre (MUHC), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Habib B, Buckeridge D, Bustillo M, Marquez SN, Thakur M, Tran T, Weir DL, Tamblyn R. Smart About Meds (SAM): a pilot randomized controlled trial of a mobile application to improve medication adherence following hospital discharge. JAMIA Open. 2021 Jul 31;4(3):ooab050. doi: 10.1093/jamiaopen/ooab050. eCollection 2021 Jul. PMID 34345805

RESULTS

PARTICIPANT FLOW:
Groups:
- SAM Intervention Group: At discharge from hospital, patients (and/or caregivers) received access to Smart About Meds (SAM), a medication management mobile application that has been developed by the McGill Clinical and Health Informatics (MCHI) Research Group.
- Usual Care Group: At discharge from hospital, patients were provided with a written discharge prescription to be filled at their community pharmacy, and may or may not have received written or verbal instructions about changes made to therapy.
Period: Overall Study
Arm/Group | SAM Intervention Group | Usual Care Group
Started | 34 | 32
Completed | 23 | 26
Not Completed | 11 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SAM Intervention Group | Usual Care Group | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54.6 [38.2 to 74.2] | 68.6 [62.1 to 76.4] | 64.6 [45.3 to 75.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 12 | 18 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Participant has caregiver [Count of Participants; unit: Participants] | 1 | 7 | 8
ED visit in 3 months prior to admission [Count of Participants; unit: Participants] | 15 | 14 | 29
Hospitalization in 3 months prior to admission [Count of Participants; unit: Participants] | 5 | 5 | 10
Number of medications prescribed at discharge [Median (Inter-Quartile Range); unit: medications] | 13.0 [8.0 to 16.0] | 15.5 [11.0 to 19.0] | 15.0 [11.0 to 18.0]
Number of medications continued at discharge [Median (Inter-Quartile Range); unit: medications] | 6.0 [4.0 to 12.0] | 11.5 [6.0 to 14.0] | 9.0 [5.0 to 13.0]
Number of medications changed at discharge [Median (Inter-Quartile Range); unit: medications] | 6.0 [4.0 to 11.0] | 7.0 [3.0 to 9.0] | 7.0 [4.0 to 10.0]
Number of new medications at discharge [Median (Inter-Quartile Range); unit: medications] | 3.0 [1.0 to 5.0] | 3.0 [1.0 to 5.0] | 3.0 [1.0 to 5.0]
Number of dose changes at discharge [Median (Inter-Quartile Range); unit: medications] | 1.0 [0.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
Number of discontinued medications at discharge [Median (Inter-Quartile Range); unit: medications] | 2.0 [0.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]

OUTCOME MEASURES:

1. Primary Outcome: Usability of the SAM App
Description: Users were observed as they used the app, following the "think aloud protocol". This involved users verbalizing their thoughts as they perform a standardized set of tasks, while being audio-recorded.A field assistant familiar with the SAM app observed and recorded users as they accessed SAM and completed the following standardized tasks: log in, peruse drug information, send the pharmacist a message, add a medication review, use the interaction checker, and use the side effect checker. User performance was observed and registered by a trained research assistant to establish if the user was able to complete the task and to determine the ease/difficulty with which the task was completed, rated in 1-to-4 scale as (1) user can do it perfectly, without any help, (2) user can do it with difficulty but without help, (3) user can do it with difficulty and help, and (4) user cannot do it.
Time Frame: At baseline, prior to hospital discharge
Population: This analysis population included 31 patients who consented to participate in the pilot and who were randomized to the intervention group and baseline and were successfully administered the questionnaire. It includes some individuals who were withdrawn from the study following randomization for various reasons (e.g. withdrew consent, discharged to a rehabilitation center, transferred to a non-study unit) and not included in other outcome analysis populations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAM Intervention Group
Number analyzed (Participants) | 31
score on a scale
  Severity scale mean, login | 1.14 (0.51)
  Severity scale mean, view drug information | 1.32 (0.74)
  Severity scale mean, send a message | 1.35 (0.65)
  Severity scale mean, review a medication | 1.81 (1.09)
  Severity scale mean, check side effects of a specific medication | 1.13 (0.45)
  Severity scale mean, check side effect profile of all medications (side effect checker) | 1.71 (0.88)
  Severity scale mean, use interaction checker | 1.17 (0.37)

2. Primary Outcome: User Acceptance of and Satisfaction With the SAM App
Description: Participants in the intervention arm completed the Technology Acceptance Model (TAM) Questionnaire 2 weeks following discharge from hospital. The questionnaire measures users' perceived ease of use and perceived usefulness of the SAM app and their intention to use the app. The TAM questionnaire is self-administered, and consists of 38 questions on a Likert scale of 1 to 7, with responses being strongly agree (7), moderately agree (6), somewhat agree (4), neutral (4), somewhat disagree (3), moderately disagree (2), and strongly disagree (1). Responses higher on the Likert scale typically reflected higher acceptance, usability, perceived usefulenss of the app, and intent to use the app from users' perspectives.
Time Frame: 2 weeks post-discharge
Population: This analysis population includes individuals who consented to participate in the pilot, were randomized to the intervention group at baseline, and who at 2 week post-discharge agreed to complete the TAM questionnaire. Only 12 of the 23 participants in the intervention group were reachable and agreed to complete the questionnaire at this point during follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAM Intervention Group
Number analyzed (Participants) | 12
score on a scale
  TAM domain: behavioral intention | 5.17 (2.12)
  TAM domain: perceived usefulness | 5.29 (2.11)
  TAM domain: subjective norm | 3.81 (1.74)
  TAM domain: relevance | 4.86 (1.78)
  TAM domain: output quality | 5.44 (1.65)
  TAM domain: result demonstrability | 5.06 (1.82)
  TAM domain: perceived ease of use | 5.65 (2.02)
  TAM domain: computer self-efficacy | 5.60 (2.00)
  TAM domain: perceived enjoyment | 5.34 (1.97)

3. Primary Outcome: Proportion of Medication Changes That Are Adhered to
Description: Pharmacy claims data from the public insurance provider will be used to identify community medications dispensed to participating patients in the 30 days following hospital discharge. These data will be compared with the patient's hospital discharge prescription to identify non-adherence to in-hospital medication changes. Non-adherence to in-hospital treatment changes in the 30-day post-discharge period will be defined as (1) failure to fill newly prescribed medications, (2) re-filling a previous prescription that was stopped at discharge, or (3) filling a previous prescription whose dosage was modified at discharge, but was dispensed post-discharge at the incorrect daily dose. For each type of medication change, the number of changes among all patients will be counted (e.g. number of newly prescribed medications among the patient population), and the number of those that were properly adhered to will then be used to calculate the proportion of medication changes that were adhered to.
Time Frame: 30 days post-discharge
Measure: Number; unit: proportion of medication changes
Arm/Group | SAM Intervention Group | Usual Care Group
Number analyzed (Participants) | 23 | 26
proportion of medication changes
  Proportion of all medication changes adhered to | 0.837 | 0.778
  Proportion of all new medications adhered to | 0.727 | 0.617
  Proportion of all dose changes adhered to | 0.909 | 0.818
  Proportion of all discontinued medications adhered to | 0.935 | 0.943

ADVERSE EVENTS:
Description: All-cause mortality, serious adverse events, and other adverse events were not monitored.
Arm/Group | SAM Intervention Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT04676165/Prot_SAP_000.pdf